CLINICAL TRIAL: NCT06076889
Title: Power Over Pain Portal: A Stepped-care Virtual Solution to Deliver Early Intervention to Canadian Youth With Chronic Pain
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Other Study IDs: REB#
Record Dates: First submitted 2023-09-13; First posted 2023-10-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Power over Pain Portal — Youth from different ages, sexes, gender, sexual orientations, races, dwelling and school/employment status will receive access to the portal for 2 months. The portal consists of self-assessment tools (bi-weekly check-ins to provide users with feedback on their mood, anxiety, pain, and sleep and guide decision making on choice of interventions), evidence-based virtual educational (pain neuroscience) and cognitive behavioural therapy (CBT) pain interventions that are delivered in a stepped care manner based on participant needs/preference.

SUMMARY:
The COVID-19 pandemic is presenting one of the greatest threats to youth mental health seen in generations. Pain is one of the most common symptoms of extreme stress in youth. In 2020, the investigators created an online "stepped-care" program called the Power over Pain Portal. Stepped care is a promising way to improve access to CP care. Stepped care tailors care based on a person's symptom severity. Like a ladder, a person must start with one type of care then "step up" or "step down" to more or less intense care depending on need. The investigators also summarized all online pain management programs for youth to find the best resources to embed into the Portal. The investigators will pilot-test the Portal with youth to ensure it can be implemented effectively and will be clinically beneficial. The investigators will recruit 100 youth with CP to use the Portal for 2 months and see how they interact with the features and if it helps to improve their pain and mental health. The investigators will include a mixture of youth who represent different ages, sexes, genders, sexual orientations, races, dwellings, and school/employment status.

ELIGIBILITY:
Inclusion Criteria:

* Experience chronic pain
* Speak and read English
* Access to Internet / Smartphone (or will be loaned study phone with data plan)
* Intend to use the portal for 2 months

Exclusion Criteria:

* Youth self-reports:
* Receiving tertiary care or are on waitlists for tertiary care paediatric chronic pain programs
* Have moderate to severe cognitive impairment that may impact their ability to understand and use the Power over Pain Portal or complete self-reported outcomes
* Have untreated major psychiatric illness (e.g., anorexia, psychosis) and/or active suicidality at the time of screening

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from a community-based sample of 100 youth with chronic pain using respondent-driven sampling (RDS), a network-based (i.e. snowball-type) method wherein a diverse group of youth with chronic pain ("seeds") provide study information to members of their social networks
  As per RDS recommendations, the "seeds" will be sociodemographically diverse, live in a variety of geographical areas, and be "high energy sociometric stars" who are committed to the study goals (i.e., our diverse youth advisory group). this strategy will seek to maximize variability in age, sex, gender, ethnicity, SES and rurality.
  This study focuses on youth marginalized by membership in racialized groups, SES as defined by neighbourhood, rural/urban status, sex and gender, and sexual orientation. Those belonging to a racialized group, living in a low SES neighbourhood, and/or rural location will be considered marginalized.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 8 weeks
  This will be assessed using the Acceptability e-Scale administered at T2 and assessed during the post-implementation qualitative interview. The minimum value is 1 and the maximum value is 5. Higher scores on the Acceptability e-Scale indicate a better outcome.
Adoption (i.e.,rate of uptake of the Power over Pain Portal) | 8 weeks
  Characterized via the user-level analytics of interactions with each feature. The benchmark will be 75% of users completing 3/4 portal assessment and accessing ≥ portal intervention.
Appropriateness (i.e., perceived fit and compatibility of the Power over Pain Portal to the needs of users) | 8 weeks
  Assessed via the post-implementation qualitative interview.
Portal Feasibility as assessed by the extent to which the Power over Pain Portal can be used as planned | 8 weeks
  Assessed using frequency counts and percentages of types/severity of problems encountered via monthly audit of technical support tickets
Portal Feasibility as assessed by the extent to which the Power over Pain Portal can be used as planned | 8 weeks
  Assessed via characterization of the severity of encountered issues on the Power over Pain portal
Fidelity | 8 weeks
  Characterized by intervention use analytics.

SECONDARY OUTCOMES:
Client outcomes | 8 weeks
  Pain intensity as assessed by the 1-item PROMIS pediatric numeric rating scale v1.0 - Pain Intensity. This maximum score on the scale is 10 and the minimum score is 0, with higher scores indicating higher levels of pain experienced by the participant. This will be administered at T1 and T2
Client outcomes | 8 weeks
  Pain interference as assessed by the the PROMIS pediatric short form v2.0 - Pain Interference 8a. The maximum score on the scale is 5 and the lowest score is 1, with higher scores indicating higher pain interference in the participant's life. This will be administered at T1 and T2.
Client outcomes | 8 weeks
  Anxiety as assessed by the the PROMIS pediatric short form v2.0 - Anxiety 8a. The maximum score on the scale is 5 and the lowest score is 1, with higher scores indicating higher levels of anxiety in the participant's life. This will be administered at T1 and T2.
Client outcomes | 8 weeks
  Depressive symptoms as assessed by the the PROMIS pediatric short form v2.0 - Depressive Symptoms 8a. The maximum score on the scale is 5 and the lowest score is 1, with higher scores indicating higher levels of depression in the participant's life. This will be administered at T1 and T2.
Client outcomes | 8 weeks
  Insomnia as assessed by the the 7-item Insomnia Severity Index. The maximum score on the scale is 4 and the lowest score is 0, with higher scores indicating more severe levels of insomnia experienced by the patient. This will be administered at T1 and T2.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada